CLINICAL TRIAL: NCT03865966
Title: Clinical Follow-up Study on Hepatitis B Virus Infection After Liver Transplantation in Children
Brief Title: Hepatitis B Virus Infection After Liver Transplantation in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qiu Li (Other)
Responsible Party: Sponsor-Investigator, Qiu Li, Principal Investigator, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 2019-24
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and liver tissue specimens。
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — No intervention

SUMMARY:
China is a highly prevalent area of hepatitis B virus（HBV） infection, with at least 75 million hepatitis B virus carriers, and 80% of primary hepatocellular carcinoma (HCC) is associated with chronic hepatitis B virus infection. Liver transplantation is currently the preferred method for end-stage liver disease such as biliary atresia and cirrhosis in children. In recent years, children's liver transplantation has developed rapidly and the number of developments has increased significantly. If there is chronic hepatitis B virus infection in the donor liver, it may cause HBV transmission, or the patient may have a low-load occult hepatitis B virus infection, and after immunosuppressive treatment, it may lead to hepatitis B virus infection after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage liver disease who require liver transplantation

Exclusion Criteria:

* Children without liver transplantation refer to children;
* Children who are unwilling to participate;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: End-stage liver disease requires liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-05 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of occult hepatitis b virus infection | 3-5 years
  Clinical follow-up testing for occult HBV infection after liver transplantation in children
The rate of overt hepatitis b virus infection | 3-5 years
  Clinical follow-up testing for overt HBV infection after liver transplantation in children

SECONDARY OUTCOMES:
The levels and changes of anti-HBs after liver transplantation | 3-5 years
  Clinical follow-up testing for HBV seromarkers after liver transplantation in children

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, Principal Investigator — Chongqing Children's Hospital of Chongqing Medical University
Locations (1):
- Chongqing Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 3-5 years